CLINICAL TRIAL: NCT07205874
Title: Early Diagnosis of Primary Biliary Cholangitis (PBC) in Patients With Positive Anti-Mitochondrial Antibodies (AMA) and Normal Alkaline Phosphatase (ALP)
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Dolores Martín Arranz, PhD, Head of department, Hospital Universitario La Paz
Other Study IDs: PI-6171
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Primary Biliary Cholangitis (PBC)
Keywords: Primary Biliary Cholangitis (PBC); Anti-Mitochondrial Antibodies (AMA); Alkaline Phosphatase (ALP)
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case patients: Patientes aged 18-80 years, with positive AMA (≥1:40 titer) and persistently normal ALP

SUMMARY:
The goal of this observational study is to achieve early diagnosis of Primary Biliary Cholangitis (PBC) in patients with positive Anti-Mitochondrial Antibodies (AMA) and Normal Alkaline Phosphatase (ALP) in adults aged 18-80 years with positive AMA and normal ALP. The main question it aims to answer is:

• Are there any predictive factors for histological PBC in patients with positive AMA and normal ALP? Participants will undergo a liver biopsy and specific blood tests if eligible based on inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Positive AMA (≥1:40 titer)
* Persistently normal ALP

Exclusion Criteria:

* Previously diagnosed with PBC, autoimmune hepatitis, or primary sclerosing cholangitis
* Under treatment with ursodeoxycholic acid, fibrates, biologics or immunosuppressants including oral steroids
* Contraindications for liver biopsy
* Concomitant debilitating disease or poor prognosis
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-80 years with positive AMA and normal ALP
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Scheuer's criteria | Just once, at enrollment
  Liver biopsy samples

SECONDARY OUTCOMES:
Enhanced Liver Fibrosis (ELF) Score | Just once, at enrollment
  Utilizes biomarkers such as hyaluronic acid, tissue inhibitor of metalloproteinase-1 (TIMP-1), and procollagen III amino-terminal peptide (PIIINP)
Fibroblast Growth Factor 19 (FGF-19) | Just once, at enrollment
  Provides insights into bile acid regulation and metabolic liver function. Quantified using enzyme-linked immunosorbent assay (ELISA)
Tumor Necrosis Factor-alpha (TNF-α) | Just once, at enrollment
  Measured via high-sensitivity ELISA to assess inflammatory status
Cytokine Profiling (Interleukin-6, -12, -23) | Just once, at enrollment
  Serum cytokine levels will be determined using multiplex immunoassays
Transforming Growth Factor-beta (TGF-β) | Just once, at enrollment
  Quantified via ELISA to evaluate its role in fibrosis and immune regulation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided